CLINICAL TRIAL: NCT05971511
Title: Current Practice for Management of Pneumothorax in Egypt
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kareem Ahmed Hosny, Dr, Assiut University
Other Study IDs: AssiuutCTS
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Pneumothorax
MeSH Terms: conditions — Pneumothorax | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire

SUMMARY:
There are standard well-known guidelines for pneumothorax management with minimal difference between societies and associations. We are investigating how much of these guidelines are actually being followed in different healthcare facilites in Egypt. This is a questionnaire that will be sent to all healthcare givers in Egypt acorss different cities and facilities with multiple choice questions presenting different case scenarios and the management options being given to the patient.

ELIGIBILITY:
Inclusion Criteria:

* being health care giver concerned with management of pneumothorax

Exclusion Criteria:

* being not concerned with management of pneumothorax

Ages: 1 Week to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare givers dealing with pneumothorax patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-27 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
Management of pneumothorax | 1 month
  Mutiole choices question to choose from

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes